CLINICAL TRIAL: NCT00930670
Title: Evaluation of the Influence of Statins and Proton Pump Inhibitors on Clopidogrel Antiplatelet Effects
Acronym: SPICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Jean-Pierre Dery, MD, MSc, Interventional Cardiologist, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SPICE
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
Keywords: ranitidine; pantoprazole; esomeprazole; omeprazole; atorvastatin; rosuvastatin; statin; clopidogrel resistance; antiplatelet therapy; coronary artery disease; percutaneous coronary intervention; stent; clopidogrel; proton pump inhibitors; drug interactions; drug resistance; genetic polymorphism
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Rosuvastatin-omeprazole (Experimental): Rosuvastatin-omeprazole
  Interventions: Drug: Rosuvastatin-omeprazole
- Rosuvastatin-pantoprazole (Experimental): Rosuvastatin 20 mg for 1 month, then rosuvastatin 20 mg and pantoprazole 40 mg for 11 months
  Interventions: Drug: Rosuvastatin-pantoprazole
- Rosuvastatin-esomeprazole (Experimental): Rosuvastatin 20 mg for 1 month, then rosuvastatin 20 mg and esomeprazole 40 mg for 11 months
  Interventions: Drug: Rosuvastatin-esomeprazole
- Rosuvastatin-ranitidine (Active Comparator): Rosuvastatin 20 mg for 1 month, then rosuvastatin 20 mg and ranitidine 300 mg for 11 months
  Interventions: Drug: Rosuvastatin-ranitidine
- Atorvastatin-omeprazole (Experimental): Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and omeprazole 20 mg for 11 months
  Interventions: Drug: Atorvastatin-omeprazole
- Atorvastatin-pantoprazole (Experimental): Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and pantoprazole 40mg for 11 months
  Interventions: Drug: Atorvastatin-pantoprazole
- Atorvastatin-esomeprazole (Experimental): Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and esomeprazole 40 mg for 11 months
  Interventions: Drug: Atorvastatin-esomeprazole
- Atorvastatin-ranitidine (Active Comparator): Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and ranitidine 300mg for 11 months
  Interventions: Drug: Atorvastatin-ranitidine

INTERVENTIONS:
Drug: Rosuvastatin-omeprazole — Rosuvastatin 20 mg for 1 month. Then rosuvastatin 20mg and omeprazole 20mg for 11 months
  Arms: Rosuvastatin-omeprazole
Drug: Rosuvastatin-pantoprazole — Rosuvastatin 20 mg for 1 month, then rosuvastatin 20 mg and pantoprazole 40 mg for 11 months
  Arms: Rosuvastatin-pantoprazole
Drug: Rosuvastatin-esomeprazole — Rosuvastatin 20 mg for 1 month, then rosuvastatin 20 mg and esomeprazole 40 mg for 11 months
  Arms: Rosuvastatin-esomeprazole
Drug: Rosuvastatin-ranitidine — Rosuvastatin 20 mg for 1 month, then rosuvastatin 20 mg and ranitidine 300mg for 11 months
  Arms: Rosuvastatin-ranitidine
Drug: Atorvastatin-omeprazole — Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and omeprazole 20 mg for 11 months
  Arms: Atorvastatin-omeprazole
Drug: Atorvastatin-pantoprazole — Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and pantoprazole 40 mg for 11 months
  Arms: Atorvastatin-pantoprazole
Drug: Atorvastatin-esomeprazole — Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and esomeprazole 40 mg for 11 months
  Arms: Atorvastatin-esomeprazole
Drug: Atorvastatin-ranitidine — Atorvastatin 80mg for 1 month, then atorvastatin 80 mg and ranitidine 300mg for 11 months
  Arms: Atorvastatin-ranitidine

SUMMARY:
There is conflicting evidence in the literature suggesting that the use of proton pump inhibitors (PPIs), and/or some statins can interfere with clopidogrel antiplatelet effect and result in adverse cardiovascular outcomes in patients treated with coronary artery stents and dual antiplatelet therapy.

The primary aim of the study is to determine the effect of various currently used PPI on platelet aggregation in patients undergoing percutaneous coronary intervention (PCI) and treated with dual antiplatelet therapy.

The secondary aim of the study is to evaluate how statins and 2C19*2 polymorphism modulate the effect of PPI on clopidogrel efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older
* Bare metal stent implantation
* Discharged with dual antiplatelet therapy for at least 60 days
* Written informed consent

Exclusion Criteria:

* Patients who do not consent to participate in the study
* Premenopausal women not using contraceptive methods or without a negative pregnancy test in the past week
* Patients treated or planned to be treated with oral anticoagulants
* Present treatment with or clear indication for treatment with a PPI or H2 antagonists
* Allergy or intolerance to study medications including ranitidine, Proton pump inhibitors, atorvastatin, rosuvastatin, aspirin and/or clopidogrel
* Patient treated with a strong CYP2C19 interacting drug
* History of a bleeding diathesis, or evidence of active abnormal bleeding within 30 days before enrollment
* History of intracranial hemorrhage or intracranial surgery in the last 3 months
* History of gastro-intestinal ulcers in the last 3 months
* Any serious illness or any condition that the investigator feels would influence the impact of this therapy on the subject
* Known platelet count < 100000/mm3 at time of enrollment or within 24 hours prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percent change in residual platelet aggregation by light transmittance aggregometry and percent change in platelet reactivity index by VASP | At 30 and 60 days

SECONDARY OUTCOMES:
Resistance to clopidogrel by light transmittance aggregometry (defined by RPA >55%), resistance to clopidogrel by vasodilator-stimulated phosphoprotein (VASP) (defined by PRI >55%) | 30 and 60 days
Prevalence and role of CYP 2C19*2 polymorphism on the effect of PPIs and statins on the antiplatelet activity of clopidogrel | 30 and 60 days
The composite of death from all causes, myocardial infarction, ischemia-driven repeat revascularization, and stroke | 30 days, 60 days and 1 year
Need to stop any antiplatelet medication for gastrointestinal bleeding or peptic ulcer disease | 30 days, 60 days and one year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Dery, MD, MHS, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Harvey A, Modak A, Dery U, Roy M, Rinfret S, Bertrand OF, Larose E, Rodes-Cabau J, Barbeau G, Gleeton O, Nguyen CM, Proulx G, Noel B, Roy L, Paradis JM, De Larochelliere R, Dery JP. Changes in CYP2C19 enzyme activity evaluated by the [(13)C]-pantoprazole breath test after co-administration of clopidogrel and proton pump inhibitors following percutaneous coronary intervention and correlation to platelet reactivity. J Breath Res. 2016 Jan 27;10(1):017104. doi: 10.1088/1752-7155/10/1/017104. PMID 26815196